CLINICAL TRIAL: NCT00735865
Title: Lid Margin And Conjunctival Microbial Flora Following Punctum Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Sarkis H. Soukiasian, M.D., Lahey Clinic, Inc.
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-049
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; Punctal Occlusion; Punctal Plugs; Tear Drainage duct blockage
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Punctal Plugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Procedure: Punctal plugs, punctal cautery
- 2 (Active Comparator)
  Interventions: Procedure: Punctal Plug, Punctal thermocauterization
- 3 (Active Comparator)
  Interventions: Procedure: Silicone plug or thermodynamic hydrophobic acrylic plug
- 4 (Active Comparator)
  Interventions: Other: Previous subjects with Punctal occlusion

INTERVENTIONS:
Procedure: Punctal plugs, punctal cautery — 25 subjects(20 silicone punctal plugs, 5 punctal cautery) The procedure will be based on clinical indication. Randomized one eye for study. Baseline cultures of lid margin & tarsal/inferior fornix conjunctiva obtained & plated according to protocol
  Arms: 1
Procedure: Punctal Plug, Punctal thermocauterization — Up to 5 subjects. Subjects in need of punctal occlusion(No preference for punctal thermocauterization or punctal occlusion by silicone plug). Randomize one eye to silicone punctal plug occlusion, the other eye to punctal thermocauterization.
  This group ONLY, cultures will be obtained of the lid margin & conjunctiva/inferior fornix of BOTH eyes
  Arms: 2
Procedure: Silicone plug or thermodynamic hydrophobic acrylic plug — Up to 5 subjects. Subjects in need of punctal occlusion(not preference for punctal occlusion by silicone plug or by the thermodynamic hydrophobic acrylic plug). Randomize one eye to silicone punctal plug occlusion, the other eye to acrylic punctal plug occlusion.
  In this group ONLY cultures will be obtained of the lid margin and conjunctiva/inferior fornix of BOTH eyes
  Arms: 3
Other: Previous subjects with Punctal occlusion — Up to 20 subjects(15 subjects with silicone punctal plug closure and 5 subjects with punctal closure by thermocauterization)Subjects who have previously had punctal occlusion who have symptoms and/or signs thought to be secondary to punctal occlusion.
  Lid margin and conjunctiva/inferior fornix of eye with greatest sign or symptoms will be cultured/plated according to standard protocol.
  Arms: 4

SUMMARY:
To determine if the types and amount of bacteria or other germs change over time after the routine procedure of blockage of tear drainage duct in the treatment of dry eye condition or other condition benefiting from a tear drainage blockage

DETAILED DESCRIPTION:
This study will investigate the impact of punctal occlusion on the ocular microbial flora. Current thought is that punctal occlusion causes retention of inflammatory mediators on the ocular surface which may produce pathology, we hypothesize that blockage of the nasolacrimal drainage system may allow colonization of the ocular surface by potentially pathogenic ubiquitous organisms (which may produce exotoxins and other biologic products) that may be responsible for signs and symptoms seen in some patients. Additionally, the presence of the silicone foreign body(punctal plug) may act as a nidus for bacterial adhesion with biofilm production (which is known to occur with Pseudomonas sp and other organisms). There would thus be a paradigm shift of our current understanding of the pathophysiology of punctal occlusion. Additionally, the choice of antimicrobials for the treatment of infections in patients with punctal occlusion may need to be modified if the microbial flora is found to be different in patients with punctal occlusion.

The ocular flora may be different inpatients with severe dry eye or other chronic pathologic conditions, which are frequent indications for punctal occlusion. However, from our retrospective review, we could not determine if there was a change in the microbial flora following plug placement with colonization with these "unusual organisms" since baseline cultures prior to punctal plug placement were not obtained.

We will try to differentiate any effect on the microbial flora caused by the silicone plug or acrylic plug(as a foreign body) versus the punctal closure by thermocautery. (Punctal thermocauterization is an alternative method of punctal closure which is 1) the preferred choice by some ophthalmologists for all their cases, or 2) when the dry eye is severe and irreversible punctal occlusion is desired or 3) if punctal plugs can not be retained due to the large size of the patients punctal). The thermodynamic hydrophobic acrylic plug(SmartPLUG) approved by the FDA for punctal occlusion with the same indications as the traditional silicone plug.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to sign Informed Consent
* Clinical indication for punctal plug insertion or punctal cautery or symptomatic patients who have previously had punctal occlusion
* Clinical indication for punctal plug removal(Partial extrusion, discomfort) increased signs of ocular irritation with punctate keratopathy, punctal inflammation).
* Able to make follow up visit schedule

Exclusion Criteria:

* Subjects without dry eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-07; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Impact of punctal occlusion on the ocular microbial flora | 1 year(3mo, 6mo, 12 mo culture/follow up visits)

CONTACTS AND LOCATIONS:
Overall Officials: Sarkis H. Soukiasian, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (2):
- United States (2):
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Lahey Clinic North, Peabody, Massachusetts